CLINICAL TRIAL: NCT00690040
Title: Single Balloon Catheter Compared With Double Balloon Catheter for Ripening of the Unfavorable Cervix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Raed Salim, MD, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0007-08-EMC
Record Dates: First submitted 2008-05-31; First posted 2008-06-04 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2013-05

CONDITIONS: Induction of Labor
Keywords: Induction of labor; Ripening; Single balloon catheter; Double balloon catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Ripening of the unfavorable cervix is done with Single balloon catheter (Foley catheter)
  Interventions: Device: Foley catheter
- 2 (Active Comparator): Ripening of the unfavorable cervix is done with double balloon catheter (Atad catheter)
  Interventions: Device: Atad catheter

INTERVENTIONS:
Device: Foley catheter — Single balloon catheter
  Arms: 1
Device: Atad catheter — Double balloon catheter
  Arms: 2

SUMMARY:
The purpose of this study is to compare between single balloon catheter and double balloon catheter for ripening the cervix among pregnant with unfavorable cervix.

ELIGIBILITY:
Inclusion Criteria:

* Induction of labor is indicated
* Gestational age between 24 - 42 weeks
* Singleton pregnancy
* Bishop score less than 7

Exclusion Criteria:

* Any contraindication for vaginal delivery
* Previous cesarean delivery
* Low lying placenta
* Rupture of membranes
* Fetal malformations incompatible with life
* intrauterine fetal death
* Amnionitis
* Genital viral infection (HIV, hepatitis C virus

  , hepatitis B virus)
* Allergy to latex

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 293 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, MD, Principal Investigator — Department of Ob/Gyn, Ha'Emek Medical Center, Afula, and Rappaport Faculty of Medicine, Technion - Israel Institute of Technology, Haifa, Israel
Locations (1):
- Department of Ob/Gyn, Ha'Emek Medical Center, Afula, Israel

REFERENCES:
- [Background] Lyndrup J, Nickelsen C, Weber T, Molnitz E, Guldbaek E. Induction of labour by balloon catheter with extra-amniotic saline infusion (BCEAS): a randomised comparison with PGE2 vaginal pessaries. Eur J Obstet Gynecol Reprod Biol. 1994 Mar 15;53(3):189-97. doi: 10.1016/0028-2243(94)90118-x. PMID 8200466
- [Background] Manabe Y, Manabe A, Takahashi A. F prostaglandin levels in amniotic fluid during balloon-induced cervical softening and labor at term. Prostaglandins. 1982 Feb;23(2):247-56. doi: 10.1016/0090-6980(82)90052-1. PMID 7079521
- [Background] Sciscione AC, McCullough H, Manley JS, Shlossman PA, Pollock M, Colmorgen GH. A prospective, randomized comparison of Foley catheter insertion versus intracervical prostaglandin E2 gel for preinduction cervical ripening. Am J Obstet Gynecol. 1999 Jan;180(1 Pt 1):55-60. doi: 10.1016/s0002-9378(99)70149-3. PMID 9914578
- [Background] James C, Peedicayil A, Seshadri L. Use of the Foley catheter as a cervical ripening agent prior to induction of labor. Int J Gynaecol Obstet. 1994 Dec;47(3):229-32. doi: 10.1016/0020-7292(94)90566-5. PMID 7705527
- [Background] St Onge RD, Connors GT. Preinduction cervical ripening: a comparison of intracervical prostaglandin E2 gel versus the Foley catheter. Am J Obstet Gynecol. 1995 Feb;172(2 Pt 1):687-90. doi: 10.1016/0002-9378(95)90594-4. PMID 7856707
- [Background] Dalui R, Suri V, Ray P, Gupta I. Comparison of extraamniotic Foley catheter and intracervical prostaglandin E gel for preinduction cervical ripening. Acta Obstet Gynecol Scand. 2005 Apr;84(4):362-7. doi: 10.1111/j.0001-6349.2005.00662.x. PMID 15762966
- [Background] Atad J, Bornstein J, Calderon I, Petrikovsky BM, Sorokin Y, Abramovici H. Nonpharmaceutical ripening of the unfavorable cervix and induction of labor by a novel double balloon device. Obstet Gynecol. 1991 Jan;77(1):146-52. PMID 1984215
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Salim R, Zafran N, Nachum Z, Garmi G, Kraiem N, Shalev E. Single-balloon compared with double-balloon catheters for induction of labor: a randomized controlled trial. Obstet Gynecol. 2011 Jul;118(1):79-86. doi: 10.1097/AOG.0b013e318220e4b7. PMID 21691166

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Balloon Catheter: Ripening of the unfavorable cervix is done with Single balloon catheter (Foley catheter)
- Double Balloon Catheter: Ripening of the unfavorable cervix is done with double balloon catheter (Atad catheter)
Period: Overall Study
Arm/Group | Single Balloon Catheter | Double Balloon Catheter
Started | 145 | 148
Completed | 145 | 148
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Balloon Catheter | Double Balloon Catheter | Total
Number analyzed (Participants) | 145 | 148 | 293
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 145 | 148 | 293
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 148 | 293
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 145 | 148 | 293

OUTCOME MEASURES:

1. Primary Outcome: Average Time in Hours From Insertion of the Catheter Until Delivery
Time Frame: At the end of the study
Measure: Mean (Standard Deviation); unit: HOURS
Arm/Group | Single Balloon Catheter | Double Balloon Catheter
Number analyzed (Participants) | 145 | 148
HOURS | 19.4 (6.0) | 19.1 (6.8)

2. Secondary Outcome: To Compare Mode of Delivery, Catheter's Side Effects and Woman's Satisfaction Between the Groups
Time Frame: At the end of the study
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Single Balloon Catheter | Double Balloon Catheter
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/148
Other Adverse Events (participants affected / at risk) | 0/145 | 0/148

LIMITATIONS AND CAVEATS:
Blinding was not performed among patients and providers. However, other than the catheter type, management was standardized. Accordingly,such unblinding is not expected to affect the objectively measured outcomeS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes